CLINICAL TRIAL: NCT01859377
Title: Evaluation and Comparison of Systemic Exposure to Ibuprofen After Single Oromucosal Versus Oral Administrations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V00498 TA 1 01; 2013-000732-96 (EudraCT Number)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ibuprofen

ARMS (2):
- Sequence 1 (Other): Test Drug (V0498 - A mg) - Reference (Ibuprofen)
  Interventions: Drug: V0498 - A mg; Drug: Ibuprofen
- Sequence 2 (Other): Reference (Ibuprofen) - Test drug(V0498 - A mg)
  Interventions: Drug: V0498 - A mg; Drug: Ibuprofen

INTERVENTIONS:
Drug: V0498 - A mg — Single oromucosal administration
Drug: Ibuprofen — Single oral administration

SUMMARY:
The purpose of this study is to evaluate the systemic exposure to ibuprofen after single oromucosal administration of the test product V0498 and single oral administration of a reference product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject aged 18 to 45 years (inclusive),
* 18.5 < or = Body Mass Index < or = 30 kg/m²,
* Non-smoker for at least 6 months
* Subject agreed to be registered in the Belgium national register "VIP Check International" for this study participation .

Exclusion Criteria:

* Positive serology for Hepatitis B Virus antigens, Hepatitis C Virus or Human Immunodeficiency Virus 1 or 2 antibodies,
* Organic disorder likely to modify absorption, distribution or elimination of the medication,
* History of sensitivity to ibuprofen or other NonSteroidal Anti-Inflammatory Drugs (NSAIDs) or to any of the excipients
* Subject who has donated blood within the past 3 months,
* Subject who has forfeited his freedom by administrative or legal award, or who is under guardianship or who has been admitted in a sanitary or social institution,
* Participation in another clinical trial in the previous month or subject still within the exclusion period of a previous clinical trial or is participating in another clinical trial,

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 11 time points up to 10h after administration
Time of Maximum Concentration | 11 time points up to 10h after administration
Area Under Curve (AUC0-72) | 11 time points up to 10h after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Liège, Belgium